CLINICAL TRIAL: NCT01304589
Title: An Open Label Trial of Milnacipran in the Treatment of Women With Provoked Vestibulodynia
Brief Title: Savella in Treatment for Provoked Vestibulodynia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Candace Brown, MSN, Pharm.D., Professor, Departments of Clinical Pharmacy, Psychiatry and Obstetrics/Gynecology, University of Tennessee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSBrown SAV-MD-18
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Vestibulodynia; Vulvodynia
Keywords: provoked vestibulodynia; vulvodynia; PVD
MeSH Terms: conditions — Vulvodynia | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milnacipran (Experimental): This was an 18-week, open-label, flexible-dose exploratory trial where eligible patients were treated with 200 mg/day of milnacipran (or the maximum tolerated dose) for a total of 12 weeks. The study design involved 3 phases: screening and baseline assessment, dose escalation and stable-dose phase. All women received 12 weeks of stable dose treatment after a 6-week dose-escalation period for a total of 18 weeks of drug exposure.
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — 6-week titration period starting at 12.5mg daily and moving up to 200mg daily (or maximum tolerated dose) for 12 weeks - total treatment period is 18 weeks
  Other Names: Savella

SUMMARY:
The primary aim of this study is to determine the efficacy of milnacipran in reducing pain in women with provoked vestibulodynia (PVD), a centrally mediated pain syndrome similar to fibromyalgia, that is characterized by severe pain in the vestibule (outer vagina). The investigators will also determine whether associated symptoms in PVD, including psychological distress, impairment of sexual function, physical function, and quality of life, are correlated with a reduction in vulvar pain.

DETAILED DESCRIPTION:
This is an 18-week, open-label, flexible-dose "proof of concept" trial where women with a diagnosis of vestibulodynia will be evaluated at baseline for eligibility. Eligible patients will be openly treated with 200 mg/d milnacipran (or the maximum tolerated dose) for a total of 12 weeks. The study design involves 4 phases: screening and washout, baseline assessment, dose escalation, and stable-dose phase (Figure 1). After completing a 2-week washout of prohibited medications, patients will enter a 2-week baseline period, where they will be trained in the use of daily diaries and the tampon test, and baseline safety and efficacy data will be recorded. Patients who continue to meet the eligibility criteria at the end of the baseline period will begin a 6-week period of dose escalation. All patients will be scheduled to receive a total of 12 weeks of stable dose treatment after the 6-week dose-escalation period for a total of 18 weeks of drug exposure.

ELIGIBILITY:
Inclusion Criteria:

1. women between 18-54 years of age,
2. 'Friedrich's Criteria' must be met (report greater than six continuous months of vulvar symptoms including insertional dyspareunia or pain to touch, demonstrate on physical exam moderate to severe tenderness to light touch, localized to the vulvar vestibule [positive Cotton Swab Test] and demonstration of variable degrees of erythema of the vestibule),
3. an average pain level of "4" or greater on the 10-point tampon test and/or an average pain level of "4" or greater on the sexual intercourse pain scale(0 = no pain at all; 10 = worse pain ever) during the 2-week screening period(see Study Parameters Section), and
4. willing to use two forms of contraception during the study.

Exclusion Criteria:

1. other vulvar conditions, including dermatoses, vulvitis, vulvar papillomatosis, and atrophic vaginitis (presence of a maturation index),
2. previous vestibulectomy,
3. active vaginal infection,
4. neuropathology, including seizure disorder or syncopal episodes,
5. pregnancy or at risk for pregnancy and not using a reliable birth control method for at least 3 months prior to entering the study,
6. breastfeeding,
7. major medical illness including chronic liver disease/hepatic impairment, renal impairment, narrow-angle glaucoma, or uncontrolled hypertension,
8. major psychiatric illness including substance abuse,
9. multiple allergies (greater than three drugs or environmental agents),
10. use of centrally-acting agents, including monoamine oxidase inhibitors, benzodiazepines, opiates, muscle relaxants, and antidepressants within 2 weeks of randomization and during the study, and
11. use of topical lidocaine, within 2 weeks of randomization and during the study, as it has shown to be an effective treatment in some women, while worsening symptoms in others. Subjects will be permitted to take acetaminophen, aspirin, or a nonsteroidal anti-inflammatory drug as rescue medication. They will be provided with a list of allowable escape medications and those which would constitute a protocol deviation.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace S Brown, PharmD, Principal Investigator — University of Tennessee
Locations (1):
- Women's Health Specialists, PLLC, Germantown, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Milnacipran: Open-label study of milnacipram. 50 to 200 milligrams orally per day. Tablets were taken in the morning during an 18-week clinical trial.
Period: Overall Study
Arm/Group | Milnacipran
Started | 31
Completed | 18
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- Milnacipram: Open-label study of milnacipram. 50 to 200 milligrams orally per day. Tablets were taken in the morning during an 18-week clinical trial.
Arm/Group | Milnacipram
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Pain Rating Index [Mean (Standard Deviation); unit: units on a scale] — The Pain Rating Index is a component of the McGill Pain Questionnaire which measures sensory and affective components of pain. "0" equals no pain to "45" equals severe pain.
  units on a scale | 20.0 (8.9)
Tampon test [Mean (Standard Deviation); unit: units on a scale] — "0" equals no pain with tampon insertion to "10" equals worse pain imaginable with tampon insertion.
  units on a scale | 5.14 (3.01)
coital pain [Mean (Standard Deviation); unit: units on a scale] — "0" equals no pain with intercourse to "10" equals worse imaginable pain with intercourse.
  units on a scale | 6.94 (2.51)
24-hour vulvar pain [Mean (Standard Deviation); unit: units on a scale] — "0" equals no vulvar pain within the last 24 hours to "10" equals worse imaginable vulvar pain within the last 24 hours.
  units on a scale | 2.09 (2.03)

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Index
Description: The Pain Rating Index is a component of the McGill Pain Questionnaire which measures sensory and affective components of pain. "0" equals no pain to "45" equals severe pain. This measure was used to measure mean values at baseline and at 18 weeks post-treatment.
Time Frame: 18 weeks
Population: 22 subjects were eligible and received study medication. Analysis population included all 22 eligible subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipram
Number analyzed (Participants) | 22
units on a scale | 12.3 (13.3)
Statistical Analysis 1: Comparison: Milnacipram; Test type: Superiority or Other; p = .001, t-test, 2 sided — A paired T-Test was calculated assuming a standard difference (d) between the 4 paired outcomes for pain of 0.60 (moderate effect size), a SD of 1 for each outcome variable and a correlation of 0.50 between each paired variable

2. Secondary Outcome: Tampon Pain
Description: "0" equals no pain with tampon insertion to "10" equals worse pain imaginable with tampon insertion. This measure was used to measure mean values at baseline and at 18 weeks post-treatment.
Time Frame: 18 weeks
Population: 22 subjects were eligible and received study medication. Analysis population includes all 22 eligible subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran
Number analyzed (Participants) | 22
units on a scale | 2.45 (2.41)
Statistical Analysis 1: Comparison: Milnacipran; Test type: Superiority or Other; p = .003, paired T-test — [p-value comment as in outcome 1, analysis 1]; Subjects completed a "tampon insertion pain" test once a week. The values were averaged and compared pre-treatment versus post-treatment

3. Secondary Outcome: Coital Pain
Description: "0" equals no pain with intercourse to "10" equals worse imaginable pain with intercourse. This measure was used to measure mean values at baseline and at 18 weeks post-treatment.
Time Frame: 18 weeks
Population: 22 subjects were assigned to study medication with 18 of the 22 subjects completing all of the study visits. Analysis population includes the 18 eligible subjects who completed all of the study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipram
Number analyzed (Participants) | 18
units on a scale | 3.43 (2.82)
Statistical Analysis 1: Comparison: Milnacipram; Test type: Superiority or Other; p = .001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: 24-hour Vulvar Pain
Description: "0" equals no vulvar pain within the last 24 hours to "10" equals worse imaginable vulvar pain within the last 24 hours. This measure was used to measure mean values at baseline and at 18 weeks post-treatment.
Time Frame: 18 weeks
Population: 22 subjects were randomized to study medication with 18 of the 22 subjects completing all of the study visits. Analysis population includes all 18 eligible subjects who completed all of the study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipram
Number analyzed (Participants) | 18
units on a scale | 0.73 (0.99)
Statistical Analysis 1: Comparison: Milnacipram; Test type: Superiority or Other; p < .001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Groups:
- Milnacipram: Crossover study
Arm/Group | Milnacipram
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 15/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipram (N=31)
nausea (Gastrointestinal disorders) | 15 (20)
headache (Nervous system disorders) | 13 (15)
hot flashes (General disorders) | 7 (9)
dizziness (Nervous system disorders) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No